CLINICAL TRIAL: NCT01460758
Title: Effectiveness of Medial Frontal Repetitive Transcranial Magnetic Stimulation With Double-Cone-Coil in Patients With Major Depression
Brief Title: Effectiveness of rTMS With Double-Cone-Coil in Patients With Major Depression
Acronym: ACDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., Principal Investigator, University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Uni-Reg-ACDC01
Record Dates: First submitted 2011-10-21; First posted 2011-10-27 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Depression
Keywords: Depression; Transcranial magnetic stimulation; rTMS; DLPFC; medial frontal cortex; anterior cingulate complex
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Medial Frontal rTMS Double-Cone-Coil (Experimental): High frequency rTMS ( Alpine Biomed Mag Pro Option) applied over medial superior frontal cortex (supplementary motor cortex) (Brodmann area 6/8),Double-Cone-water-cooled-Coil (2000 Stimuli of 10 Hz each session), 110% motor threshold.
  Interventions: Device: Medial Frontal rTMS Double-Cone-Coil
- Left DLPFC Butterfly Coil (Experimental): High frequency rTMS ( Alpine Biomed Mag Pro Option): 2000 stimuli of 10 Hz over the left DLPFC (each session), Butterfly-water-cooled-Coil, 110% motor threshold.
  Interventions: Device: Left DLPFC Butterfly Coil
- Placebo Stimulation (Sham Comparator): Sham Stimulation (Conventional butterfly-coil, angled 45°): left DLPFC continuous rTMS, 10 Hz,2000 Stimuli each session, 110% motor threshold
  Interventions: Device: Placebo Stimulation

INTERVENTIONS:
Device: Medial Frontal rTMS Double-Cone-Coil — High frequency rTMS ( Alpine Biomed Mag Pro Option) applied over medial superior frontal cortex (supplementary motor cortex) (Brodmann area 6/8),Double-Cone-water-cooled-Coil (2000 Stimuli of 10 Hz each session), 110% motor threshold.
  Arms: Medial Frontal rTMS Double-Cone-Coil
Device: Left DLPFC Butterfly Coil — High frequency rTMS ( Alpine Biomed Mag Pro Option): 2000 stimuli of 10 Hz over the left DLPFC (each session), Butterfly-water-cooled-Coil, 110% motor threshold.
  Arms: Left DLPFC Butterfly Coil
Device: Placebo Stimulation — Sham Stimulation (conventional butterfly-coil, angled 45°): left DLPFC continuous rTMS, 10 Hz, 2000 Stimuli each session, 110% motor threshold
  Arms: Placebo Stimulation

SUMMARY:
Repetitive Transcranial Magnetic Stimulation (rTMS) is used to modulate the neuronal excitability in patients with depression. In the present study the investigators will examine whether medial frontal rTMS using a double-cone-coil proves to be superior to conventional high-frequency-rTMS applied to the left-sided prefrontal cortex with a butterfly-coil.

DETAILED DESCRIPTION:
Depression is a common mental disorder that presents with depressed mood, loss of interest, feelings of guilt or low self-worth, disturbed sleep or appetite, low energy levels and poor concentration. These problems can become chronic or recurrent and lead to substantial impairments in an individual's ability to take care of his or her everyday's responsibilities, at its worst, depression can lead to suicide. Depression can be reliably diagnosed in primary care. Antidepressant medications and brief, structured forms of psychotherapy are effective for 60-80% of those affected and can be delivered in primary care.

In patients with depression the cerebral metabolism is deranged in some specific areas such as hypoexcitability in frontal cortical areas. High-frequency rTMS of the dorsolateral prefrontal cortex (DLPFC) has been investigated for the treatment of hypoexcitability disorders. Mild antidepressant effects of rTMS applied to the left sided dorsolateral prefrontal cortex (DLPFC) using a standard butterfly coil can possibly be increased by a different stimulation protocol over the medial frontal cortex using a double-cone-coil. First hints to effectiveness of this treatment arise from case reports and therefore need replication and comparability to conventional stimulation protocols. In the present study the investigators will examine whether medial frontal rTMS using a double-cone-coil proves to be more effective to conventional high-frequency-rTMS applied to the left-sided prefrontal cortex with a butterfly-coil.

ELIGIBILITY:
Inclusion Criteria:

* Episode of depression (unipolar or bipolar)( ICD-10)
* Female or male between 18 and 70 years old
* Skills to participate in all study procedures
* 18 or more points in the Hamilton rating scale or depression
* Stable antidepressant drugs
* Written informed consent

Exclusion Criteria:

* Clinically relevant unstable internal or neurological comorbidity
* Evidence of significant brain malformations or neoplasm, head injury
* Cerebral vascular events
* Neurodegenerative disorders affecting the brain or prior brain surgery
* Metal objects in and around body that can not be removed
* Pregnancy
* Alcohol or drug abuse
* Epilepsy or a pathological EEG
* Heart pacemaker
* High dose tranquillizers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-04; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in depression severity measured by the 21-item Hamilton Depression Rating Scale (Baseline versus end of treatment/ day 19) | Day 19

SECONDARY OUTCOMES:
Change in the Alertness (Baseline versus end of treatment/ day 19) | Day 19
Number of responders (response = decrease of the Hamilton Depression rating scale for at least 50%) (Baseline versus end of treatment/ day 19) | Day 19
Change in the Beck Depression Inventory (Baseline versus end of treatment/ day 19) | Day 19
Change in the Clinical Global Impression Scale (Baseline versus end of treatment/ day 19) | Day 19
Change in the Global Assessment of Functioning scale (Baseline versus end of treatment/ day 19) | Day 19
Change in the Alertness (Baseline versus follow-up I/ day 47) | Day 47
Change in the Alertness (Baseline versus follow-up II/ day 75) | Day 75
Number of responders (response = decrease of the Hamilton Depression rating scale for at least 50%) (Baseline versus follow-up I/ day 47) | Day 47
Number of responders (response = decrease of the Hamilton Depression rating scale for at least 50%) (Baseline versus follow-up II/ day 75) | Day 75
Change in the Beck Depression Inventory (Baseline versus follow-up I/ day 47) | Day 47
Change in the Beck Depression Inventory (Baseline versus follow-up II/ day 75) | Day 75
Change in the Clinical Global Impression Scale (Baseline versus follow-up I/ day 47) | Day 47
Change in the Clinical Global Impression Scale (Baseline versus follow-up II/ day 75) | Day 75
Change in the Global Assessment of Functioning scale (Baseline versus follow-up I/ day 47) | Day 47
Change in the Global Assessment of Functioning scale (Baseline versus follow-up II/ day 75) | Day 75

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, MD, Study Director — University of Regensburg - Dep. of Psychiatry; Michael Landgrebe, MD, Principal Investigator — University of Regensburg, Dpt of Psychiatry; Peter Kreuzer, MD, Principal Investigator — University of Regensburg, Dpt of Psychiatry
Locations (1):
- University of Regensburg- Dept of Psychiatry, Regensburg, Germany